CLINICAL TRIAL: NCT01227954
Title: A Phase II Trial of Hippocampal Avoidance During Whole Brain Radiotherapy for Brain Metastases
Brief Title: Avoiding the Hippocampus During Whole-Brain Radiation Therapy in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0933; CDR0000687490; NCT01366755 (obsolete NCT alias)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Cognitive/Functional Effects; Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cognitive/functional effects; tumors metastatic to brain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WBRT with Hippocampal Avoidance (Other): Whole brain radiotherapy (WBRT) with hippocampal avoidance using intensity-modulated radiation therapy (IMRT)
  Interventions: Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Radiation: intensity-modulated radiation therapy — 30 Gy in 10 fractions to the whole brain using intensity-modulated radiation therapy excluding the hippocampal avoidance area. Bilateral hippocampal contours manually generated on the fused planning MRI CT image set by the treating physician according to protocol-specified contouring instructions. Hippocampal avoidance regions generated by three-dimensionally expanding the hippocampal contours by 5 mm.
  Other Names: IMRT

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to kill tumor cells.

PURPOSE: This phase II trial is studying how well avoiding the hippocampus during whole-brain radiation therapy works in treating patients with brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate delayed recall as assessed by the Hopkins Verbal Learning Test-Revised (HVLT-R) at 4 months after hippocampal avoidance during whole-brain radiotherapy (HA-WBRT) in patients with brain metastasis.

Secondary

* Evaluate auditory and visual learning and memory, as assessed by two CogState tests (International Shopping List Test and One Card Learning Test), after HA-WBRT in these patients.
* Compare psychometric properties of the 2 CogState tests to the HVLT-R for the assessment of memory decline after HA-WBRT in these patients.
* Evaluate health-related quality of life [as assessed by the Functional Assessment of Cancer Therapy with Brain Subscale (FACT-BR) and the Barthel Index of Activities of Daily Living (ADLs)] after HA-WBRT in these patients.
* Evaluate time to radiographic progression after HA-WBRT in these patients.
* Evaluate overall survival of these patients after HA-WBR.
* Evaluate the adverse events of HA-WBR.
* Evaluate predictive biomarkers of cognitive function.

OUTLINE: This is a multicenter study.

Patients undergo 10 fractions of intensity-modulated whole-brain radiotherapy (WBRT), avoiding hippocampal (HA) regions, once daily, 5 days a week, for 2-2½ weeks.

Patients neurocognitive functions (delayed recall, auditory and visual learning, and memory) are evaluated by the Hopkins Verbal Learning Test-Revised (HVTL-R), The One Card Learning Test (OCLT), and the International Shopping List Test (ISLT) at baseline and periodically during study.

Patients may undergo serum, plasma, or whole blood collection at baseline and at 4 months after completion of HA-WBRT for correlative studies.

Patients may complete the Functional Assessment of Cancer Therapy with Brain Subscale (FACT-BR), and the Barthel Index of Activities of Daily Living (ADLs) quality-of-life questionnaires at baseline and periodically during study and follow up.

After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically or cytologically confirmed non-hematopoietic malignancy within the past 5 years

  * If histologic proof of malignancy is from > 5 years ago, then a more recent pathological confirmation is required (e.g., from systemic metastatic or brain metastasis)
  * Patients with metastasis of unknown primary tumor are permitted
* Measurable brain metastasis outside a 5-mm margin around either hippocampus on gadolinium contrast-enhanced MRI obtained within the past 30 days
* Have not been or will not be treated with stereotactic radiosurgery (SRS) or surgical resection

  * These treatment options are allowed only at relapse
* Patients who have brain metastases at initial presentation allowed and do not need to demonstrate 3 months of stable scans
* At least 1 week since open biopsy
* Karnofsky performance status 70-100%
* Fertile patients must use effective contraception
* Negative pregnancy test 2 weeks or less prior to study entry
* Patients must be English proficient, with patients who speak English as a second language eligible

EXCLUSION CRITERIA:

* Small cell lung cancer or germ cell malignancy
* Leptomeningeal metastases
* Non-small cell lung cancer-associated brain metastases with ≥ 2 organ sites of extracranial metastases
* Radiologic evidence of hydrocephalus
* Serum creatinine > 1.4 mg/dL within 30 days prior to study entry
* Pregnant or nursing
* Contraindication to MRI imaging such as implanted metal devices or foreign bodies or severe claustrophobia
* Severe, active co-morbidity including any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy
  * Uncontrolled, clinically significant cardiac arrhythmias
* Prior radiotherapy to the brain
* Plan for chemotherapy or targeted therapies during WBRT or during the subsequent 7 days

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-03; Primary Completion 2013-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minesh P. Mehta, MD, Principal Investigator — University of Maryland Medical Systems
Locations (63):
- United States (60):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Center for Cancer Care - Peoria, Peoria, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Oncology - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - NSMC Cancer Center - Peabody, Danvers, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - Nebraska Medical Center, Omaha, Nebraska
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Regional Cancer Center - Erie, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Texas Oncology, PA at Harris Center HEB, Bedford, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - Memorial Hermann Hospital - Memorial City, Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
- Canada (3):
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Gondi V, Pugh SL, Tome WA, Caine C, Corn B, Kanner A, Rowley H, Kundapur V, DeNittis A, Greenspoon JN, Konski AA, Bauman GS, Shah S, Shi W, Wendland M, Kachnic L, Mehta MP. Preservation of memory with conformal avoidance of the hippocampal neural stem-cell compartment during whole-brain radiotherapy for brain metastases (RTOG 0933): a phase II multi-institutional trial. J Clin Oncol. 2014 Dec 1;32(34):3810-6. doi: 10.1200/JCO.2014.57.2909. Epub 2014 Oct 27. PMID 25349290

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WBRT With Hippocampal Avoidance
Started | 113
Completed | 100 (Eligible subjects available for analysis)
Not Completed | 13
Not completed — Protocol Violation | 6
Not completed — No protocol treatment | 7

BASELINE CHARACTERISTICS:
Population: Eligible patients
Arm/Group | WBRT With Hippocampal Avoidance
Number analyzed (Participants) | 100
Age, Continuous [Median (Full Range); unit: years] | 61 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Delayed Recall at 4 Months as Measured by the Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: Change in Hopkins Verbal Learning Test-Revised delayed recall (HVLT_R DR) score from baseline to 4 months after the start of treatment calculated as (baseline score - 4 month score)/ baseline score. A positive change indicates a decline in function. The HVLT-R assesses verbal learning and memory. It incorporates 6 different forms, helping to mitigate practice effects of repeated administrations. Each form includes 12 nouns (targets) with 4 words drawn from 3 semantic categories, which differ across the 6 forms. Delayed recall involves recalling a list of 12 targets after a 20-minute delay. The score is the sum of the number of targets correctly recalled. Percent change calculated as 100*[(baseline score - 4 month score)/ baseline score]
Time Frame: Baseline and 4 months from start of treatment
Population: Eligible patients who started treatment and had baseline and 4 month data
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | WBRT With Hippocampal Avoidance
Number analyzed (Participants) | 42
percent change | 7.0 [-4.7 to 18.7]
Statistical Analysis 1: Comparison: WBRT With Hippocampal Avoidance; To detect a minimum relative 50% improvement leading to an absolute 15% mean relative decline (MRD) in HVLT-R DR, 51 analyzable patients were required to ensure 80% statistical power with 0.05 alpha. Assuming a death rate of 40% before 4 months (based on trial NCT00003563) and a 10% nonevaluable rate, the target sample size was 102. The target MRD was determined from NCT00003563 which demonstrated 30% MRD in HVLT-R DR score from baseline to 4 months, with a standard deviation of 41%; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percent Change at 4 Months in Auditory Learning Measured by Cogstate's International Shopping List Test (ISLT)
Description: The score is the total number of correct responses made in remembering the list on three consecutive trials in a single session. A higher score indicates a better performance. Each patient served as her or his own control, and the percent change in ISLT score from baseline to 4 months was calculated as 100*[(baseline score - 4 month score)/ baseline score].
Time Frame: Baseline and 4 months from start of treatment
Population: Eligible patients who started treatment and had baseline and 4 month data
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | WBRT With Hippocampal Avoidance
Number analyzed (Participants) | 34
percent change | 18.0 [5.5 to 30.5]

3. Secondary Outcome: Percent Change at 4 Months in Visual Learning Measured by Cogstate's One Card Learning Test (OCLT)
Description: The score is the arcsine of the square root of the proportion of correct responses. A higher score indicates a better performance. Each patient served as her or his own control, and the percent change in OCLT score from baseline to 4 months was calculated as 100*[(baseline score - 4 month score)/ baseline score].
Time Frame: Baseline and 4 months from start of treatment
Population: Eligible patients who started treatment and had baseline and 4 month data
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | WBRT With Hippocampal Avoidance
Number analyzed (Participants) | 34
percent change | -8 [-16.9 to 0.9]

4. Secondary Outcome: Quality of Life as Measured by the Functional Assessment of Cancer Therapy-Brain (FACT-Br)
Description: The FACT-Br is a 19-item self-report instrument designed to measure multidimensional quality of life in patients with brain cancer. It is to be administered with the FACT-General. The FACT-G is a validated, 27-item measure where a higher score represents higher QOL. In addition to a total QOL score, subscale scores for physical, functional, social and emotional well-being are produced. There are 5 responses options, 0=Not a lot to 4=Very much. All subscale items are added together, multiplied by the number of items in the subscale, then divided by the number of items answered to obtain subscale totals. Scores range 0-108 for FACT-G total, 0-28 for physical, social, functional subscales, 0-24 for emotional subscale, 0-76 for brain subscale. Certain items must be reversed before it is added by subtracting the response from 4. Subscale requires >= 50% of items to be completed while the overall response rate must be > 80%. If items are missing, the subscale scores can be prorated.
Time Frame: Baseline and 4 months from start of treatment
Population: Eligible patients who started treatment and completed at least one FACT-Br assessment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | WBRT With Hippocampal Avoidance
Number analyzed (Participants) | 80
units on a scale
  Baseline: number analyzed (Participants) | 78
  Baseline | 121.25 [74 to 158]
  2 month: number analyzed (Participants) | 48
  2 month | 111.94 [85 to 158]
  4 month: number analyzed (Participants) | 37
  4 month | 115 [81 to 159]
  6 month: number analyzed (Participants) | 25
  6 month | 126.22 [90.83 to 159]
Statistical Analysis 1: Comparison: WBRT With Hippocampal Avoidance; A general linear fixed effects model was run with FACT-Br total score (baseline, 2, 4, 6 mo. from end of treatment) as outcome of interest. Explanatory variables: Age (>= 60 vs. <60), primary site (lung,breast,colon each vs. other), neurologic function status (no vs. some symptoms), and recursive partitioning analysis class (RPA) (I vs. II). Explanatory variables are reported separately and only if in the final model (p< 0.10, except time forced in the model.). Intercept is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable in the final model is reported separately
Statistical Analysis 2: Comparison: WBRT With Hippocampal Avoidance; A general linear fixed effects model was run with FACT-Br total score (baseline, 2, 4, 6 mo. from end of treatment) as outcome of interest. Explanatory variables in the model: Age (>= 60 vs. <60), primary site (lung,breast,colon each vs. other), neurologic function status (no vs. some symptoms), and RPA class(I vs. II). Explanatory variables are reported separately and only if they are in the final model (p< 0.10, except time forced in the model.). Time is reported here; Test type: Superiority; p = 0.1961, Mixed Models Analysis; Each explanatory variable in the final model is reported separately
Statistical Analysis 3: Comparison: WBRT With Hippocampal Avoidance; A general linear fixed effects model was run with FACT-Br total score (baseline, 2, 4, 6 mo. from end of treatment) as outcome of interest. Explanatory variables in the model: Age (>= 60 vs. <60), primary site (lung,breast,colon each vs. other), neurologic function status (no vs. some symptoms), and RPA class(I vs. II). Explanatory variables are reported separately and only if they are in the final model (p< 0.10, except time forced in the model.). Primary site (lung) is reported here; Test type: Superiority; p = 0.0715, Mixed Models Analysis; Each explanatory variable in the final model is reported separately
Statistical Analysis 4: Comparison: WBRT With Hippocampal Avoidance; A general linear fixed effects model with FACT-Br total score (baseline, 2, 4, 6 mo. from end of treatment) as outcome of interest. Explanatory variables in the model: Age (>= 60 vs. <60), primary site (lung,breast,colon each vs. other), neurologic function status (no vs. some symptoms), and RPA class(I vs. II). Explanatory variables are reported separately and only if they are in the final model (p< 0.10, except time forced in the model.). Neurologic status (no symptoms) is reported here; Test type: Superiority; p = 0.0554, Mixed Models Analysis; Each explanatory variable in the final model is reported separately

5. Secondary Outcome: Quality of Life as Measured by the Barthel Index of Activities of Daily Living (ADL)
Description: The Barthel Index of Activities of Daily Living (ADL) is a 10-item assessment. Patient scores on the ADL range from 0 to 20 with lower scores indicating declining functional status.
Time Frame: Baseline and 4 months from start of treatment
Population: Eligible patients who started treatment and completed at least one ADL assessment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | WBRT With Hippocampal Avoidance
Number analyzed (Participants) | 81
units on a scale
  Baseline: number analyzed (Participants) | 80
  Baseline | 20 [10 to 21]
  2 month: number analyzed (Participants) | 49
  2 month | 20 [5 to 20]
  4 month: number analyzed (Participants) | 38
  4 month | 20 [7 to 20]
  6 month: number analyzed (Participants) | 24
  6 month | 20 [13 to 20]
Statistical Analysis 1: Comparison: WBRT With Hippocampal Avoidance; A general linear fixed effects model was run with ADL (baseline, 2, 4, 6 mo. from end of treatment) as outcome of interest. Explanatory variables in the model: Age (>= 60 vs. <60), primary site (lung,breast,colon each vs. other), neurologic function status (no vs. some symptoms), and RPA class(I vs. II). Explanatory variables are reported separately and only if they are in the final model (p< 0.10, except time forced in the model.). Intercept is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable in the final model is reported separately
Statistical Analysis 2: Comparison: WBRT With Hippocampal Avoidance; A general linear fixed effects model was run with ADL (baseline, 2, 4, 6 mo. from end of treatment) as outcome of interest. Explanatory variables in the model: Age (>= 60 vs. <60), primary site (lung,breast,colon each vs. other), neurologic function status (no vs. some symptoms), and RPA class(I vs. II). Explanatory variables are reported separately and only if they are in the final model (p< 0.10, except time forced in the model.). Time is reported here; Test type: Superiority; p = 0.1579, Mixed Models Analysis; Each explanatory variable in the final model is reported separately
Statistical Analysis 3: Comparison: WBRT With Hippocampal Avoidance; A general linear fixed effects model was run with ADL (baseline, 2, 4, 6 mo. from end of treatment) as outcome of interest. Explanatory variables in the model: Age (>= 60 vs. <60), primary site (lung,breast,colon each vs. other), neurologic function status (no vs. some symptoms), and RPA class(I vs. II). Explanatory variables are reported separately and only if they are in the final model (p< 0.10, except time forced in the model.). Neurologic function status (some symptoms) is reported here; Test type: Superiority; p = 0.0559, Mixed Models Analysis; Each explanatory variable in the final model is reported separately
Statistical Analysis 4: Comparison: WBRT With Hippocampal Avoidance; A general linear fixed effects model was run with ADL (baseline, 2, 4, 6 mo. from end of treatment) as outcome of interest. Explanatory variables in the model: Age (>= 60 vs. <60), primary site (lung,breast,colon each vs. other), neurologic function status (no vs. some symptoms), and RPA class(I vs. II). Explanatory variables are reported separately and only if they are in the final model (p< 0.10, except time forced in the model.). Age (>= 60) is reported here; Test type: Superiority; p = 0.0749, Mixed Models Analysis; Each explanatory variable in the final model is reported separately

6. Secondary Outcome: Overall Survival
Description: Overall survival was measured from registration to the date of death or last known follow-up (censored). Kaplan-Meier estimator was used to median survival time and 95% confidence interval.
Time Frame: Analysis occurs after all patients have been on study for at least 4 months. (Patients are followed from registration to death or study termination whichever occurs first.)
Population: Eligible patients who started study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | WBRT With Hippocampal Avoidance
Number analyzed (Participants) | 96
months | 6.8 [4.8 to 10.9]

7. Secondary Outcome: Progression-free Survival
Description: Progression (radiographic) is defined as an increase in perpendicular bidimensional tumor area (at lease 50% for lesions < 1cm, at least 25% for lesions >=1cm) for any of the 1-3 tracked brain metastases, or the appearance of any new brain metastasis on a follow-up MRI. Progression-free survival was calculated instead of time to progression. Progression-free survival time was measured from registration to the date of progression, death, or last known follow-up (censored). The Kaplan-Meier method used to determine median time (along with 95% confidence intervals).
Time Frame: as for outcome 6
Population: Eligible patients who started study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | WBRT With Hippocampal Avoidance
Number analyzed (Participants) | 96
months | 5.9 [4.7 to 8.4]

8. Secondary Outcome: The Frequency of Patients With Grade 3 and Higher Adverse Events (AE) Related to Treatment
Description: For each patient the highest grade adverse event related to treatment was calculated. Those with their highest grade of 3 or higher were counted. Adverse events are graded using CTCAE v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE
Time Frame: From start of treatment to 12 months from start of treatment
Population: Eligible patients who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | WBRT With Hippocampal Avoidance
Number analyzed (Participants) | 96
Participants | 2

9. Secondary Outcome: ApoE4 Genotype and Other Potentially Predictive Biomarkers of Cognitive Function
Description: Per the protocol, the feasibility of the proposed translational studies were to be assessed following completion of accrual and sample collection. The decision was made not to pursue this outcome measure. No assays were performed and no data were collected for this Outcome Measure
Time Frame: Baseline and 4 months from start of treatment
Arm/Group | WBRT With Hippocampal Avoidance
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Eligible patients with adverse event data are included. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | WBRT With Hippocampal Avoidance
Serious Adverse Events (participants affected / at risk) | 13/96
Other Adverse Events (participants affected / at risk) | 46/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WBRT With Hippocampal Avoidance (N=96)
Anemia (Blood and lymphatic system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Colonic perforation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 2
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cognitive disturbance (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | WBRT With Hippocampal Avoidance (N=96)
Blurred vision (Eye disorders) | 8
Constipation (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 34
Gait disturbance (General disorders) | 7
Weight loss (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 13
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 17
Memory impairment (Nervous system disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.